CLINICAL TRIAL: NCT00593723
Title: IMRT Tomotherapy for Esophagus Cancer: A Phase I Feasibility Study in Non-Operative Patients
Brief Title: IMRT Tomotherapy for Esophagus Cancer
Acronym: IMRT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-1070 / 201105499
Record Dates: First submitted 2008-01-02; First posted 2008-01-15 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: Esophagus Cancer
Keywords: IMRT
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IMRT + Concurrent chemotherapy (Experimental): 180 cGy daily fractions to a total dose of 5400 cGy to PTV1 and 200 cGy daily fractions to a total dose of 6000 cGy to PTV2. Once a day, five days a week, for approximately 6 weeks.
  Planned chemotherapy: cisplatin (75 mg/m2) day 1 and 5-FU (1000 mg/m2) days 1-4 on weeks 1, 5, 10, and 14 of therapy. Please note that drug regimens and doses may vary and will be at the discretion of the medical oncologist.
  Interventions: Radiation: IMRT

INTERVENTIONS:
Radiation: IMRT

SUMMARY:
Concurrent chemotherapy and radiation therapy are the standard of care for inoperable patients with esophagus cancer. Unfortunately, the 5-year survival of 20% for this population is quite low. Methods to intensify radiation therapy delivery without increasing local toxicities are needed. Intensity modulated radiation therapy (IMRT) is an advanced method of delivering external beam radiation that may minimize the volume of normal tissue irradiated to high dose and thus decrease the risk of normal tissue toxicity. The proposed study will prospectively test whether IMRT is tolerable for delivering IMRT doses of 60 Gy for patients with esophagus cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18
* Karnofsky Performance Status of >= 60
* TNM Stages T1-4, N0-3, M0
* Pathologic confirmation of esophagus cancer
* Evaluation by medical oncologist determines that the patient is medically fit for concurrent chemotherapy
* Evaluation by surgeon determines that patient is unresectable

Exclusion Criteria:

* Age < 18
* Karnofsky Performance Status < 60
* Radiographic or pathologic evidence of distant metastatic disease (classified as M1b in AJCC staging manual)
* Prior radiation therapy to the thorax or upper abdomen, preventing definitive radiation therapy.
* Pregnant or lactating, if female.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2006-12; Primary Completion 2014-01 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The study will evaluate the feasibility of using helical tomotherapy to deliver IMRT in patients with unresectable esophagus cancer. | One year after protocol registration
  The study will be deemed infeasible if one or more of the following results occur:
  * 15% of patients experience any grade 4 acute toxicity judged to be related to his/her external radiation treatment
    * within 1 year of protocol registration, >15% of patients develop any grade 4 late toxicity judged to be related to his/her external radiation treatment
    * within 1 year of protocol registration, any patient dies from causes judged to be related to his/her external beam radiation treatment

SECONDARY OUTCOMES:
Evaluate local recurrence rates | Until patient progressive disease or death
  6 weeks after therapy, every 3 months for first two years post therapy, every 6 months for years 3, 4, and 5 post therapy, and then annually.
Evaluate disease-free survival rates | Until patient progressive disease or death
  6 weeks after therapy, every 3 months for first two years post therapy, every 6 months for years 3, 4, and 5 post therapy, and then annually.
Evaluate regional recurrence rates | Until patient progressive disease or death
  6 weeks after therapy, every 3 months for first two years post therapy, every 6 months for years 3, 4, and 5 post therapy, and then annually.
Evaluate distant recurrence rates | Until patient progressive disease or death
  6 weeks after therapy, every 3 months for first two years post therapy, every 6 months for years 3, 4, and 5 post therapy, and then annually.
Evaluate overall survival rates | Until patient progressive disease or death
  6 weeks after therapy, every 3 months for first two years post therapy, every 6 months for years 3, 4, and 5 post therapy, and then annually.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Bradley, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu